CLINICAL TRIAL: NCT05960422
Title: Effects of Adding Adductor Canal Block to Popliteal Sciatic Nerve Block in Hallux Valgus Correction Operations
Brief Title: Popliteal Sciatic Nerve Block and Adductor Canal Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Ezgi POLAT, Principal Investigator, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EzgiPOLAT
Record Dates: First submitted 2023-07-17; First posted 2023-07-25 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Popliteal Sciatic Nerve Block; Adductor Canal Block
Keywords: Popliteal sciatic block, adductor canal block

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Popliteal Sciatic Nerve Block (Active Comparator): Patients are in the group undergoing popliteal sciatic block
  Interventions: Procedure: Popliteal Sciatic Nerve Block
- Adductor Canal Block (Active Comparator): Patients are in the group undergoing popliteal sciatic block + adductor canal block
  Interventions: Procedure: Adductor canal block

INTERVENTIONS:
Procedure: Popliteal Sciatic Nerve Block — Patients undergoing popliteal sciatic block, the side where the procedure would be performed in the prone position was sterilized after appropriate antisepsis. After visualizing the popliteal artery in the popliteal fossa with the probe it was advanced proximally in a horizontal and minimally lateral position to determine the point of separation of the tibial and peroneal nerves from the sciatic nerve. Subcutaneous local anesthesia was applied at this point after the skin, and the stimulator needle was advanced towards the sciatic nerve in an in-plane approach, passing through the skin and subcutaneous tissue, and then the nerve stimulator was opened up to 1 mA. After observing motor movement in the foot, the stimulator was reduced to 0.3-0.5 mA, and after observing motor movements for duration of 0.1 ms, 10 ml of 0.5% bupivacaine + 10 ml of 2% prilocaine were administered to the target tissue
  Arms: Popliteal Sciatic Nerve Block
Procedure: Adductor canal block — Patients in the group undergoing popliteal sciatic block + adductor canal block, with the extremity to be blocked slightly externally rotated, the anterior part of the thigh was prepared with the necessary antiseptic procedures while the patient was in the supine position. Using an ultrasound probe, the femoral artery was visualized by advancing the ultrasound probe distally, and the saphenous nerve was identified just lateral to the femoral artery, beneath the sartorius muscle. At the junction of the sartorius muscle and vastus medialis, 10 ml of 0.5% bupivacaine + 10 ml of 2% prilocaine were applied to the periphery of the saphenous nerve. Subsequently, the patient was turned prone, and a popliteal sciatic block was performed.
  Arms: Adductor Canal Block

SUMMARY:
The goal of this observational study is to determine the effect of adding adductor canal block to popliteal sciatic nerve block on patient-surgeon satisfaction, intraoperative sedation need, tourniquet pain, return time of motor block, and postoperative pain in patients undergoing hallux valgus correction surgery. The main question it aims to answer are:

* Does peroperative pain decrease?
* Do patient-surgeon satisfaction increase? The patients were divided into two groups, the Popliteal Sciatic Block (PSB) group, and the Popliteal Sciatic Block + Adductor Canal Block (PSB + ACB) group.

DETAILED DESCRIPTION:
Patients were randomly assigned into 2 groups as popliteal sciatic nerve block (Group PSB), popliteal sciatic nerve + adductor canal block (Group PSB + ACB). In this study, 52 patients scheduled for hallux valgus correction operations, in the American Society of Anesthesiologists I-III groups, between the ages of 18-80, were enrolled. Study was planned as a prospective, randomized and controlled trial. All patients were perfomed PSB with 10 ml 0.5% bupivacaine and 10 ml 2% prilocaine in the prone position, using ultrasonography and nerve stimulator. 10 ml of 0.5% bupivacaine and 10 ml of 2% prilocaine were administered to the patients in the ACB + PSB group in the supine position, in addition to PSB. Patients with coagulopathy, infection at the region site of regional blockade, allergy of local anesthetic drugs, peripheral neuropathy and neurogenic disorders affecting the lower extremities, peripheral artery disease, mental retardation and those who did not give consent to study were excluded. All patients were sedated with 1-2 mg midazolam and 50 µg fentanyl. After the blocks were performed , sensory -motor block onset time, surgery-tourniquet time, tourniquet pain, motor block time, pain onset time, first analgesic administration time (NPRS≥4) and analgesic administered were recorded. Anesthesiologists evaluating these data were blinded to group distribution .

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 80
* American Society of Anesthesiologists ASA I-III

Exclusion Criteria:

* Patients with coagulopathy
* Patient with wounds or infections in the region
* Patient with allergies to local anesthetic drugs
* Patient with significantly impaired peripheral neuropathy and neurogenic disorders affecting the lower extremity
* Patient with peripheral arterial disease
* Patient with mental retardation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | Postoperative 24 hours
  The Numeric Pain Rating Scale (NPRS). Between 1-10. The low values mean low pain and a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ezgi Polat, Principal Investigator — İstanbul Medeniyet University
Locations (1):
- Istanbul Medeniyet University Faculty of Medicine Department of Anesthesiology and Reanimation, Istanbul, Kadikoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No